CLINICAL TRIAL: NCT04471493
Title: Real Time Surveillance of Pediatric Infectious Diseases in French Ambulatory Care: PARI Study
Brief Title: Pediatric and Ambulatory Research in Infectious Diseases
Acronym: PARI
Status: Recruiting | Type: Observational
Sponsor: Association Clinique Thérapeutique Infantile du val de Marne (Other)
Collaborators: AFPA (Association Française de Pédiatrie Ambulatoire) (Unknown); GlaxoSmithKline (Industry); Sanofi (Industry); Pfizer (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: ACT0116
Record Dates: First submitted 2020-07-08; First posted 2020-07-15 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Otitis; Bronchiolitis; Influenza; Pharyngitis; Varicella; Pneumonia; Gastroenteritis
Keywords: Vaccination; Antibiotic treatment; Point of care test; automated data extraction; network
MeSH Terms: conditions — Otitis; Bronchiolitis; Influenza, Human; Pharyngitis; Chickenpox; Pneumonia; Gastroenteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Many ambulatory networks are mainly based on diagnoses made by first-line physicians not specifically trained to join the network. Here we aim to set up a surveillance network on pediatric infectious diseases with an investment in teaching with specific trainings of participating pediatricians, increasing in use of point of care tests, and automated data extraction from the computers of the pediatricians.

DETAILED DESCRIPTION:
107 pediatricians among the 1400 members of the French ambulatory pediatric association, AFPA (Association Française de Pédiatrie Ambulatoire) were involved in this survey.To belong to the PARI network, pediatricians have to use the same software, Axi5-Infansoft (developed by CompuGroup Medical, Nanterre, France) for electronic medical record of children. The pediatricians were trained to the use of point of care tests and to the infectious diagnoses (otitis, pharyngitis, varicella, bronchiolitis, influenza, pneumonia, etc..). The study population consisted of all children under 16 years of age from the patient population for which an infectious disease was diagnosed.

ELIGIBILITY:
Inclusion Criteria:

* Children under 16 years of age with at least one infectious disease among:
* pharyngitis
* otitis
* pneumonia
* influenza
* bronchiolitisz
* varicella
* gastroenteritis
* enterovirus disease
* bordetella pertussis disease
* using the same same software, Axi5-Infansoft (developed by CompuGroup Medical, Nanterre, France)

Exclusion Criteria:

* parental refusal

Ages: 1 Day to 16 Years | Sex: All
Age Groups: Child
Study Population: Children under 16 years with infectious disease
Sampling Method: Probability Sample
Enrollment: 400000 (Estimated)
Dates: Start 2017-06-26 (Actual); Primary Completion 2030-06-27 (Estimated); Study Completion 2030-08-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the number of infectious diseases | 5 years
  proportion of children under 16 years, with infectious disease

SECONDARY OUTCOMES:
Evaluation of the use of point of care tests | 5 years
  Proportion of use of point of care tests and positivity rate according to the infectious diseases
Evaluation of the antibiotic treatments | 5 years
  Proportion of each antibiotic treatments according to the infectious diseases

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cohen, Study Director — Association Clinique et Thérapeutique Infantile du Val de Marne
Locations (1):
- AFPA, Créteil, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cohen R, Bechet S, Gelbert N, Frandji B, Vie Le Sage F, Thiebault G, Kochert F, Cahn-Sellem F, Werner A, Ouldali N, Levy C. New Approach to the Surveillance of Pediatric Infectious Diseases From Ambulatory Pediatricians in the Digital Era. Pediatr Infect Dis J. 2021 Jul 1;40(7):674-680. doi: 10.1097/INF.0000000000003116. PMID 33657594
- See also: New Approach to the Surveillance of Pediatric Infectious Diseases From Ambulatory Pediatricians in the Digital Era — https://pubmed.ncbi.nlm.nih.gov/33657594/
- See also: Trends in pediatric ambulatory community acquired infections before and during COVID-19 pandemic: A prospective multicentric surveillance study in France — https://pubmed.ncbi.nlm.nih.gov/36034052/